CLINICAL TRIAL: NCT02078921
Title: The Effects of Inorganic Nitrate on Cardiac Muscle: Physiology, Pharmacology and Therapeutic Potential in Patients Suffering From Angina
Brief Title: The Effects of Inorganic Nitrate on Cardiac Muscle in Angina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/077/11
Record Dates: First submitted 2014-02-04; First posted 2014-03-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — sodium nitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Inorganic Nitrate
  Interventions: Drug: Sodium Nitrate
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Nitrate
  Arms: Treatment
Drug: Placebo
  Arms: placebo

SUMMARY:
Previous studies have shown that interventions which modestly increase blood nitrite_ improve skeletal muscle function on exercise while sparing oxygen, and have been also shown to open up the blood flow during periods of oxygen deprivation. Inorganic nitrate in the diet is absorbed into the bloodstream, concentrated and reduced by bacteria in the mouth to nitrite, which is then absorbed into the bloodstream. .

The purpose of this study is to look at the effects of oral inorganic nitrate supplementation on clinical markers of heart ischaemia and the frequency of angina.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over with chronic stable angina (≥2 months duration).

Inclusion Criteria Following screening visit:

* A positive exercise ECG (1mmSTD at J+0.08 seconds) on a modified Bruce protocol treadmill exercise test.
* A positive dobutamine stress echocardiogram,
* and/or a positive myocardial perfusion scan (MPI),
* and/or a positive coronary angiogram.

Exclusion Criteria:

* Unable to do exercise test
* Women of child bearing potential
* If of a racial origin at risk of glucose-6-phosphate dehydrogenase (G6PD) deficiency, G6PD will be excluded prior to inclusion in the study
* Resting STD>=1mm
* NYHA 3 or 4 HF or LVEF<45%
* Myocardial infarction or revascularisation within the last two months
* Left bundle branch block (LBBB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to 1mm ST depression | 12 weeks
  The primary outcome is to assess whether oral nitrate treatment increase the time to 1mm ST depression on a modified Bruce protocol exercise test

SECONDARY OUTCOMES:
Onset of chest pain | 12 weeks
  Time to onset of chest pain on a modified Bruce protocol exercise test
Change in TDI systolic peak velocity | 12 weeks
  Change in Tissue Doppler Imaging (TDI) systolic peak velocity in ischaemic wall segments
Angina frequency | 12 weeks
  Angina frequency
GTN use frequency | 12 weeks
  GTN use frequency
Questionnaire Score | 12 weeks
  Modified Seattle Angina Questionnaire Score
Nitrate/Nitrite | 12 weeks
  Measurements of Nitrate and Nitrite in plasma
Metabolic, inflammatory and angiogenic plasma markers | 12 weeks
  Measurements of metabolic, inflammatory and angiogenic markers in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Research facility, University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Schwarz K, Singh S, Parasuraman SK, Rudd A, Shepstone L, Feelisch M, Minnion M, Ahmad S, Madhani M, Horowitz J, Dawson DK, Frenneaux MP. Inorganic Nitrate in Angina Study: A Randomized Double-Blind Placebo-Controlled Trial. J Am Heart Assoc. 2017 Sep 8;6(9):e006478. doi: 10.1161/JAHA.117.006478. PMID 28887315
- [Derived] Schwarz K, Singh S, Parasuraman SK, Bruce M, Shepstone L, Feelisch M, Minnion M, Ahmad S, Horowitz J, Dawson DK, Frenneaux MP. A randomized double-blind placebo-controlled crossover trial of sodium nitrate in patients with stable angina INAS. Future Cardiol. 2016 Nov;12(6):617-626. doi: 10.2217/fca-2016-0026. Epub 2016 Oct 12. PMID 27730819